CLINICAL TRIAL: NCT02199002
Title: Acid Pocket: Different Position and Chemical Content Between Healthy Volunteers and GERD Patients
Brief Title: Acid Pocket: Position and Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Guy Boeckxstaens, MD, PhD, KU Leuven
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S55731
Record Dates: First submitted 2014-07-17; First posted 2014-07-24 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: GERD - PPI Responders; GERD - PPI Non-responders; Barrett Esophagus; Healthy Volunteers
Keywords: acid pocket; GERD; Barrett
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- healthy volunteers (Other): healthy volunteers (no gastric complains)
  Interventions: Device: multi-pH-impedance manometry catheter
- PPI responders (Other): proven reflux, good symptom relief upon PPI therapy
  Interventions: Device: multi-pH-impedance manometry catheter
- PPI non-responders (Other): proven reflux disease, poor symptom control (less then 50% symptom reduction) upon PPI therapy (2x40mg omeprazole)
  Interventions: Device: multi-pH-impedance manometry catheter
- Barrett - no dysplasia (Other): proven barrett with no dysplasia on biopsies
  Interventions: Device: multi-pH-impedance manometry catheter
- barrett - high grade dysplasia (Other): proven barrett with high grade dysplasia on biopsies
  Interventions: Device: multi-pH-impedance manometry catheter

INTERVENTIONS:
Device: multi-pH-impedance manometry catheter — a special catheter will be placed in the esophagus of all study groups. Measurment of pH, impedance and pressure will be performed.

SUMMARY:
Gastroesophageal reflux disease (GERD) is a very common condition affecting up to 30% of adults. To date, therapy consists of powerful acid suppression with proton pump inhibitors (PPI). Nevertheless, only 60-70% of GERD patients report complete symptom relief with this therapy. As the mechanisms underlying symptom perception in PPI resistant patients are not fully understood, there is currently no adequate therapy available.

It is becoming increasingly clear that reflux, especially in the postprandial period, occurs from a reservoir of acid floating on top of the meal: the so-called "acid pocket". In this study, we aim to investigate further the acid pocket by determining its exact position and chemical contents between healthy volunteers, GERD patient who respond well and bad to PPI therapy and GERD patients with barrett's esophagus.

DETAILED DESCRIPTION:
A costume made multi-pH-impedance manometry catheter will be placed in the esophagus and clipped to the Z-line. Patients then will be given a standardized meal and the position of the acid pocket will be measured. After two hours the pocket will be aspirated through a gastric catheter. Then, patients will be allowed to return home and the study will be continued for another 22 hours.

The special catheter will be removed at the end of the study. Collected acid pockets will be used to analyze content and perform permeability experiments.

Data of the 24-hour experiment will be used to evaluate the position of the acid pocket and number of reflux episodes.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* older than 18 years
* fit to criteria of 'study population' (HV, PPI responder, PPI non-responder, Barrett)

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-07; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
acid pocket position | participants will be followed for 24 hours
  Acid position will be determined relatively to the lower esophageal sfincter. Differences in position between healthy volunteers, PPI responders, PPI non-responders and patients with barrett esophagus will be evaluated

SECONDARY OUTCOMES:
number of reflux episodes | 24 hours
  number of reflux episodes will be counted and compared between the different groups.

OTHER OUTCOMES:
acid pocket contents | 1 year
  after collection of all acid pocket, pockets will be processed to determine it's exact chemical content.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boeckxstaens, MD, PhD, Principal Investigator — Catholic University Leuven
Locations (1):
- Catholic University Leuven, Leuven, Belgium